CLINICAL TRIAL: NCT00223899
Title: A Phase 1, Multi-Center, Open-Label, Dose-Escalation Trial to Evaluate the Safety of Intratumoral VCL-IM01 Followed by Electroporation in Metastatic Melanoma
Brief Title: A Trial to Evaluate the Safety of Intratumoral VCL-IM01 Followed by Electroporation in Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM01-101
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; Electroporation; IL-2
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): IL-2-encoding plasmid formulated in phosphate-buffered saline at 0.5 mg/mL, 1.5 mg/mL, and 5.0 mg/mL (VCL-IM01) intratumorally injected and followed by electroporation with Inovio MedPulser® 1.0 cm array with needles up to 3 cm long (one 6-pulse cycle per tumor).
  Interventions: Genetic: VCL-IM01 (encoding IL-2) with Electroporation

INTERVENTIONS:
Genetic: VCL-IM01 (encoding IL-2) with Electroporation — IL-2-encoding plasmid formulated in phosphate-buffered saline at 0.5 mg/mL, 1.5 mg/mL, and 5.0 mg/mL (VCL-IM01) intratumorally injected and followed by electroporation with Inovio MedPulser® 1.0 cm array with needles up to 3 cm long (one 6-pulse cycle per tumor).

SUMMARY:
To evaluate the safety of intratumorally injected VCL-IM01 at doses of 0.5 mg (1 tumor), 1.5 mg (1 tumor), 5 mg (1 tumor), 10 mg (2 tumors, 5 mg per tumor) and 15 mg (3 tumors, 5 mg per tumor) followed by electroporation.

DETAILED DESCRIPTION:
Eligible subjects will receive intratumoral injections of VCL-IM01 followed by electroporation of the injected tumor(s).

Subjects will be enrolled to receive one course of treatment. A course of treatment is two cycles, each cycle consisting of four weekly injection/electroporation administrations followed by an observation period of two weeks.

Subjects' tumors will be evaluated at Screening, at the end of Cycle 2, and at six months (Week 26) from the initial drug administration.

ELIGIBILITY:
Inclusion Criteria - Key criteria include:

* Confirmed recurrent metastatic melanoma
* Tumor(s) to be treated must be at least 1 cm by 1 cm, and be accessible to treatment
* Able to carry out normal daily activities and light work without assistance
* Not currently receiving chemotherapy or immunotherapy
* Normal blood chemistries and blood cell counts (elevation of LDH to less than or equal to 1.5 times normal is allowed)
* Able and willing to give informed consent.

Exclusion Criteria - Key criteria include:

* History of brain tumors (resected or stereotactically treated is allowed)
* History of liver tumors
* Subjects whose melanoma can be cured by surgery
* Pregnant
* Subjects with electronic pacemakers, defibrillators, or any other implanted electronic device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety of intratumorally injected VCL-IM01 followed by electroporation in subjects with recurrent metastatic melanoma | After all subjects have been enrolled

SECONDARY OUTCOMES:
Overall response rate, duration of response, treated tumor response rate, assessment of injected tumor(s) for induration, inflammation, and erythema, and serum levels of IL-2. | After all subjects have been enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri D. Kharkevitch, MD, PhD, Study Director — Vical
Locations (4):
- United States (4):
  - Location #2, Mobile, Alabama
  - Location #3, Denver, Colorado
  - Location #1, Chicago, Illinois
  - Location #4, Montclair, New Jersey